CLINICAL TRIAL: NCT00430560
Title: Work Activity Augmented by Cognitive Rehabilitation: Continuation and Follow-up
Brief Title: Work Activity Augmented by Cognitive Rehabilitation for Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2356-R; MDB0003
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: work therapy; cognitive rehabilitation; schizophrenia; schizoaffective disorder; treatment outcome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): work therapy
  Interventions: Procedure: work therapy; Behavioral: work therapy
- 2 (Experimental): work therapy plus cognitive remediation
  Interventions: Behavioral: cognitive rehabilitation

INTERVENTIONS:
Behavioral: cognitive rehabilitation — computer training
  Other Names: computer training
  Arms: 2
Procedure: work therapy — opportunity to work in carefully supervised hospital job
  Other Names: IWT
  Arms: 1
Behavioral: work therapy — work therapy
  Arms: 1

SUMMARY:
This research investigates the benefits of productive activity and cognitive rehabilitation for patients with schizophrenia. Key questions are:

1. does cognitive rehabilitation plus work activity produce better outcomes than work activity alone?
2. Is cognitive rehabilitation more helpful for individuals with moderate or greater cognitive impairment than for individuals without such impairment?
3. Does cognitive rehabilitation reduce the dropout rate and increase participation in work activity for cognitively impaired subjects?
4. What features of cognitive rehabilitation are most important for clinical and rehabilitation outcomes?

DETAILED DESCRIPTION:
This is a randomized, matching study in which subjects are stratified by degree of cognitive impairment, then randomly assigned to one of two conditions: Work Services Only vs. Work Services plus cognitive rehabilitation. Longitudinal analysis of work activity, work performance, symptoms, quality of life, cognitive function and service utilization are made.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia or schizoaffective disorder

Exclusion Criteria:

* change in psychiatric medications or housing within 30 days of study intake
* episode of drug abuse within 30 days of study intake
* GAF score 30 or less
* known neurological disease or developmental disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2000-10; Primary Completion 2005-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Neuropsychological test performance | data collection completed

SECONDARY OUTCOMES:
Hours of productive activity | data collection completed
Hours worked | data collection completed
Quality of life | data collection completed
Psychiatric symptoms | data collection completed

CONTACTS AND LOCATIONS:
Overall Officials: Morris D Bell, Ph.D., Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Background] Wexler BE, Bell MD. Cognitive remediation and vocational rehabilitation for schizophrenia. Schizophr Bull. 2005 Oct;31(4):931-41. doi: 10.1093/schbul/sbi038. Epub 2005 Aug 3. PMID 16079390
- [Result] Bell M, Bryson G, Wexler BE. Cognitive remediation of working memory deficits: durability of training effects in severely impaired and less severely impaired schizophrenia. Acta Psychiatr Scand. 2003 Aug;108(2):101-9. doi: 10.1034/j.1600-0447.2003.00090.x. PMID 12823166
- [Result] Bell M, Bryson G, Greig T, Corcoran C, Wexler BE. Neurocognitive enhancement therapy with work therapy: effects on neuropsychological test performance. Arch Gen Psychiatry. 2001 Aug;58(8):763-8. doi: 10.1001/archpsyc.58.8.763. PMID 11483142
- [Result] Fiszdon JM, Cardenas AS, Bryson GJ, Bell MD. Predictors of remediation success on a trained memory task. J Nerv Ment Dis. 2005 Sep;193(9):602-8. doi: 10.1097/01.nmd.0000177790.23311.ba. PMID 16131943
- [Result] Fiszdon JM, Whelahan H, Bryson GJ, Wexler BE, Bell MD. Cognitive training of verbal memory using a dichotic listening paradigm: impact on symptoms and cognition. Acta Psychiatr Scand. 2005 Sep;112(3):187-93. doi: 10.1111/j.1600-0447.2005.00565.x. PMID 16095473
- [Result] Bell MD, Fiszdon JM, Greig TC, Bryson GJ. Can older people with schizophrenia benefit from work rehabilitation? J Nerv Ment Dis. 2005 May;193(5):293-301. doi: 10.1097/01.nmd.0000161688.47164.71. PMID 15870612
- [Result] Bell MD, Bryson GJ, Greig TC, Fiszdon JM, Wexler BE. Neurocognitive enhancement therapy with work therapy: Productivity outcomes at 6- and 12-month follow-ups. J Rehabil Res Dev. 2005 Nov-Dec;42(6):829-38. doi: 10.1682/jrrd.2005.03.0061. PMID 16680620
- [Result] Fiszdon JM, Choi J, Bryson GJ, Bell MD. Impact of intellectual status on response to cognitive task training in patients with schizophrenia. Schizophr Res. 2006 Oct;87(1-3):261-9. doi: 10.1016/j.schres.2006.04.011. Epub 2006 Jun 5. PMID 16737798
- [Result] Bell MD, Fiszdon J, Bryson G, Wexler BE. Effects of neurocognitive enhancement therapy in schizophrenia: normalisation of memory performance. Cogn Neuropsychiatry. 2004 Aug;9(3):199-211. doi: 10.1080/13546800344000084. PMID 16571581